CLINICAL TRIAL: NCT01094145
Title: Deep Brain Stimulation of the Nucleus Basalis Meynert to Treat Cognitive Deficits in Light to Moderate Alzheimer's Disease
Brief Title: Deep Brain Stimulation (DBS) of the Nucleus Basalis Meynert (NBM) to Treat Cognitive Deficits in Light to Moderate Alzheimer's Disease
Acronym: MeynD-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Jens Kuhn, Prof. Dr. Jens Kuhn, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UK-09157
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Alzheimer Disease
Keywords: (light to moderate)
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Sham Comparator): Stimulator setting is OFF
  Interventions: Other: Deep brain stimulation
- Deep Brain Stimulation (Active Comparator): Stimulator setting is ON
  Interventions: Other: Deep brain stimulation

INTERVENTIONS:
Other: Deep brain stimulation — DBS in the Nucleus basalis Meynert

SUMMARY:
In the study at hand, six patients with light to moderate Alzheimer's disease will be enrolled and implanted with bilateral electrodes in the nucleus basalis Meynert.

DETAILED DESCRIPTION:
In the study at hand, six patients with light to moderate Alzheimer's disease will be enrolled and implanted with bilateral electrodes in the nucleus basalis Meynert. The stereotactic implantation of the electrodes will be guided by computerized tomography (CT) and magnetic resonance tomography (MRT).

Basically, even though deep brain stimulation is an invasive method, there are only few side effects. Surgical risks correspond with the risk of DBS in morbus Parkinson or other movement disorders (0,4-6%).

After the baseline examination, the patients will be implanted with the electrodes; accordingly all follow-ups are accomplished postoperative. From the second week after the operation, the conventional stimulation takes place as a doubleblind, randomized change between ON and OFF periods. Modifications of the stimulation parameter to obtain the best possible result are possible.

Throughout the one-year observation-period, the patients will be followed closely to monitor the effects of DBS on their cognitive abilities, psychopathological well being, the quality of life, praxie and nutritional condition using standardized neurological and psychiatric rating scales.

ELIGIBILITY:
Inclusion Criteria:

* German speaking male/female subjects
* age:60-80
* AD assessed by DSM-IV, ICD-10 and NINCDS-ADRDA-Scale
* no Lewy-Body-dementia or other form of dementia
* MMST >18 and <26
* stable psychopharmacological medication
* no psychotic symptoms, no suicidal tendency
* education for at least 8 years
* written informed consent of the patient
* consent of at least two family members
* no contraindication regarding PET-examination
* no contraindication regarding anesthesia or stereotactic operation

Exclusion Criteria:

* legal accommodation
* clinical co-morbidity
* contraindication of MRT examination
* psychotic symptoms last six months
* aggressive behavior or suicidal tendency
* verbal IQ <85
* stereotactic operation in previous history
* neoplastic neurological diseases
* serious organic disease

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
cognitive improvement | one- year
  improving cognitive outcome parameters assessed by a series of standardized neuropsychological tests

SECONDARY OUTCOMES:
determination of the optimal stimulation parameter | one year

CONTACTS AND LOCATIONS:
Overall Officials: Volker Sturm, MD, Principal Investigator — University of Cologne; Jens Kuhn, MD, Principal Investigator — University of Cologne; H. J. Freund, Prof. Dr. med., Principal Investigator — Stellvertretender Leiter der Klinischen Prüfung Institut für Neurowissenschaften und Medizin (INM-7) Forschungszentrum Jülich
Locations (1):
- Uni-Klinik Köln AöR, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Baldermann JC, Schuller T, Huys D, Becker I, Timmermann L, Jessen F, Visser-Vandewalle V, Kuhn J. Deep Brain Stimulation for Tourette-Syndrome: A Systematic Review and Meta-Analysis. Brain Stimul. 2016 Mar-Apr;9(2):296-304. doi: 10.1016/j.brs.2015.11.005. Epub 2015 Dec 29. PMID 26827109